CLINICAL TRIAL: NCT00947947
Title: Enhancing Message Design in Tailored, Computerized HIV/STI Interventions
Brief Title: Computerized HIV/Sexually Transmitted Disease (STD) Prevention Program
Acronym: TIPSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH077507 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: condom use; HIV prevention; African American; Behavioral intervention; HIV Seronegativity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention media condition (Experimental): Received a stage tailored DVD-based intervention
  Interventions: Behavioral: Tailored Information Program for Safer Sex
- standard of care (Placebo Comparator): received only clinical standard of care
  Interventions: Behavioral: Tailored Information Program for Safer Sex

INTERVENTIONS:
Behavioral: Tailored Information Program for Safer Sex — Health communication intervention delivered on a laptop computer to increase positive perceptions of condoms and increase skills to use condoms.
  Other Names: Computerized health intervention

SUMMARY:
The purpose of the current study is to test a computerized HIV/STD prevention program with heterosexual African Americans. The hypothesis is that those exposed to the program will increase their correct and consistent use of condoms compared to those not exposed to the program.

DETAILED DESCRIPTION:
The proposed study will involve the development and pilot testing of an interactive computerized tailored intervention program for HIV/STI prevention among at-risk heterosexually active African-American STI clinic patients, aged 18-29. The Attitude-Social-Influence Efficacy (ASE) model will serve as a conceptual foundation for the intervention and tailored feedback, which will assess and give feedback to participants separately for main/steady and other/casual partners. Individual modules will be developed for key theoretical concepts and subsequently tied together into an integrated system. The tailored feedback will additionally be enhanced by crafting intervention messages to be high in message sensation value and by developing interactive intervention activities for skill-building, which will be guided by both Social Cognitive Theory and skills training principles. The computerized intervention will be developed and guided using data collected from the target audience to ensure an empirically-based approach to tailoring. The intervention will also be developed with input from the target audience in order to maximize the appropriateness and persuasiveness of the feedback and the program, including interactive components. The final year of the project will entail a pilot test of the intervention in order to gather preliminary data on the acceptability and efficacy of such an intervention for increasing safer sexual behaviors among at-risk heterosexually active African-Americans.

The specific aims of the study are: 1) to develop tailored feedback on HIV/STI prevention based on the ASE model, including condom attitudes, social influences, self-efficacy including communication / negotiation skills, partner and behavioral risk, correct condom use, and condom stages of change; 2) to enhance the delivery of the tailored messages using sensation-seeking targeting (SENTAR) and skill-building using interactive activities guided by Social Cognitive Theory (SCT) and skills training principles; 3) to tie the individual theoretical modules together and develop a computerized intervention program for HIV/STI prevention, which provides tailored risk reduction messages to participants based upon an assessment of participant characteristics; 4) to develop empirically sound cutpoints, specific to the target audience, to guide the message tailoring; and 5) in a wait-list control group design, to pilot test the intervention for acceptability and efficacy in increasing condom use with main and casual partners among at-risk heterosexually active African-Americans, relative to a "usual care" comparison condition.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Aged 18-29
* Heterosexually active in past 3 months
* NOT knowingly HIV positive
* Not pregnant or planning on becoming pregnant/impregnating partner in next 3 months
* Client of the STI clinic where study is being conducted
* Not currently enrolled in another condom study at the clinic

Exclusion Criteria:

* None

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Condom use with main and casual sexual partners | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crosby, Ph.D., Principal Investigator — Department of Communication, University of Kentucky; Seth M. Noar, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Specialty Clinic, Louisville Metro Health Department, Louisville, Kentucky, United States